CLINICAL TRIAL: NCT01138397
Title: Immunogenicity and Safety of the Influenza Vaccine (Split Virion, Inactivated), Northern Hemisphere 2010-2011 Formulation (Intradermal Route)
Brief Title: Immunogenicity and Safety of a Vaccine Against Influenza (2010-2011 Northern Hemisphere Season, Intradermal Route)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID34; 2009-017688-40 (EudraCT Number); UTN: U1111-1112-2795 (Other: WHO)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine; Influenza virus; Intradermal
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Participants at 18 to 59 years of age
  Interventions: Biological: Influenza virus vaccine (split virion, inactivated)
- Group 2 (Experimental): Participants at 60 years of age or older
  Interventions: Biological: Influenza virus vaccine (split virion, inactivated)

INTERVENTIONS:
Biological: Influenza virus vaccine (split virion, inactivated) — 0.1 mL, Intradermal
  Arms: Group 1
Biological: Influenza virus vaccine (split virion, inactivated) — 0.1 mL, Intradermal
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the new formulation of the influenza vaccine for the 2010-2011 Northern Hemisphere (NH) season in terms of immunogenicity and safety in the corresponding population and to check its compliance with the Committee for Proprietary Medicinal Products (CPMP) Note for Guidance (NfG) CPMP/BWP/214/96

Objectives:

* To evaluate compliance, in terms of immunogenicity, of the corresponding strength of the intradermal (ID) influenza vaccine NH 2010-2011 formulation with the requirements of the CPMP NfG CPMP/BWP/214/96.
* To describe the safety of the corresponding strength of the ID influenza vaccine, NH 2010-2011 formulation.

DETAILED DESCRIPTION:
Each participant will receive a dose of their assigned vaccine on Day 0 and will be followed up for 21 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 years or over on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination

Exclusion Criteria :

* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination
* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* History of pandemic H1N1 influenza vaccination
* History of clinically or laboratory confirmed pandemic H1N1 influenza infection
* History of influenza vaccination within the previous 6 months (other than pandemic H1N1 influenza vaccine)
* Receipt of an adjuvanted influenza vaccine in a clinical trial within the previous 12 months
* Known or suspected congenital or acquired immunodeficiency, resulting for example from:

  * End-stage renal disease requiring dialysis
  * Active neoplastic disease or active hematologic malignancy
  * Receipt of immunosuppressive therapy or other immune-modifying drugs such as, but not limited to: anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 3 weeks following the trial vaccination
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Information concerning the immunogenicity of the Influenza virus vaccine (Split Virion, Inactivated), Northern Hemisphere 2010-2011 Formulation. | 21 days post-vaccination
Information concerning the safety (solicited and unsolicited adverse events) of the Influenza virus vaccine (Split Virion, Inactivated), Northern Hemisphere 2010-2011 Formulation. | 21 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Belgium (2):
  - Antwerp
  - Leuven

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com